CLINICAL TRIAL: NCT05866354
Title: An Open-Label, Phase 1 Trial to Evaluate Pharmacokinetics of Tisotumab Vedotin in Chinese Subjects With Metastatic or Recurrent Solid Malignancies
Brief Title: To Evaluate Pharmacokinetics of Tisotumab Vedotin in Chinese Subjects With Metastatic or Recurrent Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zai Lab (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Zai Lab (Hong Kong), Ltd. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZL-1309-002
Record Dates: First submitted 2023-04-27; First posted 2023-05-19 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Solid Malignancies
Keywords: Metastatic or Recurrent Solid Malignancies
MeSH Terms: conditions — Neoplasm Metastasis | interventions — tisotumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Tisotumab Vedotin — Tisotumab vedotin is an antibody-drug conjugate (ADC) targeting tissue factor (TF), a protein aberrantly expressed in a wide number of solid tumors including cervical cancer.

SUMMARY:
The goal of this clinical trial is to test in Chinese Subjects with Metastatic or Recurrent Solid Malignancies. The main questions it aims to answer are:

* How is the PK of tisotumab vedotin?
* How is the immunogenicity of tisotumab vedotin?
* How is the safety and tolerability of tisotumab vedotin?
* How is the clinical efficacy of tisotumab vedotin? Participants will receive 2.0 mg/kg tisotumab vedotin (up to a maximum of 200 mg in subjects ≥ 100 kg) as a 30-minute IV infusion 1Q3W with the aim to characterize the PK profiles and to evaluate immunogenicity, safety, and tolerability of tisotumab vedotin in the Chinese population.

Subjects will receive study treatment until disease progression or any other discontinuation criteria are met, whichever occurs first. Subjects will undergo an end of treatment (EOT) visit 30 days (± 5 days) after the last dose of study treatment or within 7 days after treatment discontinuation has been decided, whichever occurs later.

DETAILED DESCRIPTION:
This is an open-label, phase 1, PK trial of intravenous tisotumab vedotin in Chinese subjects with recurrent or metastatic solid tumors who have failed on previous standard systemic therapy. The screening period will be up to 28 days, after which eligible subjects will receive 2.0 mg/kg tisotumab vedotin (up to a maximum of 200 mg in subjects ≥ 100 kg) as a 30-minute IV infusion 1Q3W with the aim to characterize the PK profiles and to evaluate immunogenicity, safety, and tolerability of tisotumab vedotin in the Chinese population.

Subjects will receive study treatment until disease progression or any other discontinuation criteria are met, whichever occurs first. Subjects will undergo an end of treatment (EOT) visit 30 days (± 5 days) after the last dose of study treatment or within 7 days after treatment discontinuation has been decided, whichever occurs later.

Blood samples for the assessment of tisotumab vedotin concentrations and antidrug antibody (ADA) will be drawn in accordance with the PK and ADA collection schedule. Three different PK analytes will be measured: 1) tisotumab vedotin (conjugated antibody only), 2) total antibody (ie, conjugated and unconjugated antibody), and 3) free MMAE. PK parameters to be estimated will include, but are not limited to, AUC, Cmax, time to maximum concentration (Tmax), apparent terminal half-life (t1/2), and trough concentration (Ctrough).

Safety and tolerability will be evaluated based on TEAEs, clinical safety assessments and clinical laboratory assessments. Ocular AEs are a known safety risk of tisotumab vedotin treatment. Therefore, the eye care plan will be implemented for all subjects enrolled in this trial.

Efficacy assessments will include confirmed ORR assessed by the investigator, primarily based on the enhanced computed tomography (CT) or magnetic resonance imaging (MRI) scans performed at protocol-specified time points. The RECIST v1.1 criteria will be used for response evaluation. After discontinuation of study treatment, tumor assessments may or may not be performed at the discretion of the investigator.

At the end of study (EOS), sponsor will ensure provision of continued tisotumab vedotin to subjects with clinical benefit defined as stable disease (SD) or better, until criteria of treatment discontinuation are met.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Must sign an informed consent form (ICF) .
3. Must have recurrent or metastatic solid tumors and have failed on previous standard systemic therapy.
4. Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. Has life expectancy of at least 3 months.
6. Must demonstrate acceptable screening laboratory values.
7. Female subjects must agree not to breastfeed or donate ova. A male subject who is sexually active with a female partner of reproductive potential and has not had a vasectomy must agree to use a barrier method of birth control (eg, condom with spermicide), and all men must also not donate sperm during the trial and for 6 months after receiving the last dose of tisotumab vedotin.
8. Any other toxicity caused by previous treatment should have recovered to ≤ CTCAE grade 1 or baseline level, except ≤ CTCAE grade 2 alopecia.

Exclusion Criteria:

1. Has clinically significant bleeding issues or risks:
2. Has cardiovascular issues or risks:
3. Central nervous system (CNS): any history of intracerebral arteriovenous malformation, cerebral aneurysm, or stroke (transient ischemic attack > 1 month prior to screening is allowed).
4. Ophthalmological: active ocular surface disease or a history of cicatricial conjunctivitis or inflammatory conditions that predispose to cicatrizing conjunctivitis (eg, Wagner syndrome, atopic keratoconjunctivitis, autoimmune disease affecting the eyes), and subjects with penetrating ocular transplants are ineligible. Cataracts alone is not an exclusion criterion.
5. Surgery/procedures: major surgery within 4 weeks or minor surgery within 7 days prior to the first study treatment administration.
6. Peripheral neuropathy ≥ grade 2.
7. Any prior treatment with MMAE-derived drugs.
8. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (dose exceeding 10 mg daily of prednisone or equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of tisotumab vedotin.
9. Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject (eg, compromise well-being) or that could prevent, limit, or confound the protocol-specified assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2023-11-02 (Actual)

PRIMARY OUTCOMES:
PK parameter AUC of tisotumab vedotin | At the end of Cycle 3 (each cycle is 21 days) of the last ongoing patient, about 1 year.
  To assess PK of tisotumab vedotin.PK parameters to be estimated will include area under the concentration-time curve (AUC).
PK parameter Cmax of tisotumab vedotin | At the end of Cycle 3 (each cycle is 21 days) of the last ongoing patient, about 1 year.
  To assess PK of tisotumab vedotin.PK parameters to be estimated will include maximum concentration (Cmax).
PK parameter Tmax of tisotumab vedotin | At the end of Cycle 3 (each cycle is 21 days) of the last ongoing patient, about 1 year.
  To assess PK of tisotumab vedotin.PK parameters to be estimated will include time to maximum concentration (Tmax).
PK parameter t 1/2 of tisotumab vedotin | At the end of Cycle 3 (each cycle is 21 days) of the last ongoing patient, about 1 year.
  To assess PK of tisotumab vedotin.PK parameters to be estimated will include apparent terminal half-life (t 1/2).
PK parameter C trough of tisotumab vedotin | At the end of Cycle 3 (each cycle is 21 days) of the last ongoing patient, about 1 year.
  To assess PK of tisotumab vedotin.PK parameters to be estimated will include trough concentration (C trough).

SECONDARY OUTCOMES:
Immunogenicity of tisotumab vedotin. | At the end of Cycle 3 (each cycle is 21 days) of the last ongoing patient, about 1 year.
  Anti-drug antibodies (ADAs) against tisotumab vedotin.
Treatment-emergent adverse events (TEAEs) of tisotumab vedotin. | Through study completion, an average of 1 year.
  A TEAE is defined as a newly occurring or worsening AE from the first dose of study treatment to 30 days after the last dose of study treatment or initiation of new antitumor activities, whichever occurs first.

OTHER OUTCOMES:
Objective response rate (ORR) of tisotumab vedotin. | Through study completion, an average of 1 year.
  Confirmed objective response rate (ORR) assessed by the investigator per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Rutie Yin, Dr, Principal Investigator — West China Second University Hospital; Guiling Li, Dr, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology; Bingzhong Zhang, Dr, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Qing Wen, Dr, Principal Investigator — Jinan Central Hospital; Meili Sun, Dr, Principal Investigator — Jinan Central Hospital; Jianhua Shi, Dr, Principal Investigator — Linyi Cancer Hospital; Dongqing Lv, Dr, Principal Investigator — Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University; Tienan Yi, Dr, Principal Investigator — Xiangyang Central Hospital
Locations (1):
- Jinan Central Hospital, Jinan, Shangdong, China

IPD SHARING:
Plan to Share IPD: No
When the study close， the IPD will share to other researchers per the requirement from Zailab.